CLINICAL TRIAL: NCT06344507
Title: Iconographic Registry of Pancreatobiliary Endoscopy Procedures
Acronym: TAILOR-EUS
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Giorgio Arcidiacono, MD, Associated Professor UniSR, IRCCS San Raffaele
Other Study IDs: TAILOR-EUS
Record Dates: First submitted 2024-03-21; First posted 2024-04-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Neoplasm; Cancer of Pancreas; Pancreatitis; Neuroendocrine Tumors
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the TAILOR-EUS study (Iconographic Registry of Bilio-Pancreatic Endoscopic Ultrasound Procedures) is to establish a clinical registry comprising images and videos generated during endoscopic procedures conducted for the investigation of pancreatic diseases (PD). The study will compile historical, pathological, and imaging data from approximately 12,000 patients (2,000 retrospectively and 10,000 prospectively) who underwent endoscopic ultrasound procedures for inflammatory pancreatic conditions (e.g., acute, recurrent, chronic pancreatitis), autoimmune bilio-pancreatic diseases (e.g., autoimmune pancreatitis), neoplastic bilio-pancreatic conditions, and screenings for individuals at high risk of developing such diseases at the Bilio-Pancreatic Endoscopy and Endoscopic Ultrasound Unit of the IRCCS San Raffaele Hospital between 2000 and 2027.

Participants have undergone or will undergo the standard diagnostic pathway appropriate for their conditions as part of routine clinical practice. All instrumental examinations and endoscopic ultrasound procedures are integral to the standard diagnostic and therapeutic approach for pancreatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed diagnosis of inflammatory pancreatic disease (e.g., acute, recurrent, or chronic pancreatitis) or autoimmune bilio-pancreatic disease (e.g., autoimmune pancreatitis) or bilio-pancreatic neoplastic disease, necessitating an endoscopic ultrasonography procedure.
* Age over 18 years.
* Ability to provide informed consent.

Exclusion Criteria:

* Pregnancy and breastfeeding status.
* Contraindications to the endoscopic ultrasonography procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 12,000 patients who, between 2000 and 2027, underwent endoscopic ultrasound procedures at the Bilio-Pancreatic Endoscopy and Endoscopic Ultrasound Unit of the IRCCS San Raffaele Hospital for suspected diagnoses (based on clinical and/or diagnostic evaluations suggesting a potential diagnosis of one of the diseases listed below) and/or confirmed diseases (verified by histological and/or radiological reports when histological diagnosis was not possible).
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Registry for images and videos | Through study completion, an average of 5 years
  Establishment of a registry for images and videos captured during Endoscopic Ultrasonography (EUS) procedures, aimed at enhancing clinical data collection to improve patient diagnoses and advance the quality of Clinical Pathways for pancreatic diseases. The future goal of this initiative is to identify potential characteristics that could enhance the diagnostic yield of this technique and predict patient outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy